CLINICAL TRIAL: NCT00377884
Title: Serologic Based Molecular Characterization of Bone-healing After Cementless Total Hip Arthroplasty
Brief Title: Serologic Characterization of Bone-healing
Status: Withdrawn | Type: Observational
Why Stopped: Lack of patients, lack of funding for analysis
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: CCBR Clinical Research Center, Aalborg, Denmark (Unknown)
Responsible Party: Northern Orthopaedic Division, Orthopaedic Research Unit, Aarhus University - Aalborg Hospital, Denmark
Other Study IDs: ON-04-018-MBL
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Arthritis
Keywords: THA
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Investigation of serologic bone markers in patients undergoing hip arthroplasty

DETAILED DESCRIPTION:
Investigation of serologic bone markers in patients undergoing hip arthroplasty. Measured by frequent blood- and urine samples pre-operative and during the first post-operative year.

ELIGIBILITY:
Inclusion Criteria:

* Ages 40-80 years

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients planned for cementless THR for OA in the hip
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mogens B Laursen, MD, Phd, Principal Investigator — Northern Orthopaedic Division
Locations (2):
- Denmark (2):
  - Northern Orthopaedic Division, Aalborg, Northern Jutland
  - Aalborg University Hospital, Aalborg